CLINICAL TRIAL: NCT06751524
Title: Botensilimab and Balstilimab Expanded Access Program
Brief Title: Expanded Access Program (EAP) Designed to Provide Access to Botensilimab and Balstilimab Before Regulatory Approval
Status: Available | Type: Expanded Access
Sponsor: Agenus Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: BOTBAL EAP
Record Dates: First submitted 2024-12-20; First posted 2024-12-30 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Colorectal Cancer (CRC); Pancreatic Cancer; Non-Small Cell Lung Cancer (NSCLC); Hepatocellular Carcinoma (HCC); Melanoma; Sarcoma; Ovarian Cancer; Prostate Cancer
Keywords: Compassionate Use; Early Access; Expanded Access; Managed Access; Pre-approval Access; Special Access; Named Patient Program (NPP)
MeSH Terms: conditions — Colorectal Neoplasms; Pancreatic Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Hepatocellular; Melanoma; Sarcoma; Ovarian Neoplasms; Prostatic Neoplasms | interventions — balstilimab

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Botensilimab — Administered via an intravenous (IV) infusion of Botensilimab + Balstilimab combination (BOT+BAL).
  Other Names: AGEN 1181
Drug: Balstililmab — Administered via an IV infusion of Botensilimab + Balstilimab combination (BOT+BAL).
  Other Names: AGEN 2034

SUMMARY:
This is an expanded access program (EAP) designed to provide access to Botensilimab and Balstilimab prior to drug registration by the applicable local regulatory agency. A medical doctor must decide whether the potential benefit outweighs the risk of receiving an investigational therapy based on the individual patient's medical history and program eligibility criteria.

DETAILED DESCRIPTION:
This EAP is available for indications where there is reasonable scientific basis for use. Availability will depend on territory eligibility.

ELIGIBILITY:
Key Inclusion Criteria:

* The patient's disease is serious or life-threatening.
* The patient has undergone appropriate standard treatments; there are no comparable or satisfactory alternative treatments for the disease or condition; the treatment is adjunct to an existing treatment option, and the treatment is not medically contra-indicated.
* Sufficient efficacy and safety evidence exists to make a benefit-risk analysis consistent with this policy and the potential patient benefit justifies any potential risks of treatment.
* Sufficient clinical data are available to identify an appropriate dose and treatment duration.
* The patient's treating physician and qualified medical personnel at Agenus agree there is sufficient evidence to assume the potential benefit to the patient justifies potential risks.
* The patient is not eligible for participation in an ongoing clinical trial of the investigational medicine, including lack of access due to geographic limitations.
* Expanded Access will not adversely impact any clinical development program, in particular, the conduct of a pivotal clinical trial that is required for regulatory approval.
* The request must be made by the patient's treating physician.

Note: Other defined Inclusion/Exclusion criteria may apply.

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Agenus Inc.

REFERENCES:
- See also: Agenus Medical Affairs — https://agenusbio.com/medical-affairs/
- See also: Agenus Clinical Trials — https://agenusbio.com/clinical-trials/
- See also: Agenus Access to Investigational Medicines Policy — https://agenusbio.com/access-to-investigational-medicines-policy